CLINICAL TRIAL: NCT01176331
Title: Outcomes of 20 and 23-gauge Combined Transconjunctival Pars Plana Vitrectomy
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Other Study IDs: KOU-8487358664
Record Dates: First submitted 2010-08-03; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-07

CONDITIONS: Vitrectomy

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- vitrectomy
  Interventions: Procedure: 20 and 23 gauge pars plana vitrectomy

INTERVENTIONS:
Procedure: 20 and 23 gauge pars plana vitrectomy

SUMMARY:
In a retrospective study, a combined 20 and 23-gauge pars plana vitrectomy procedure was performed in 21 eyes for various indications and proposed as a transition procedure to 23-gauge transconjunctival vitrectomy. Through use of combination of procedures postoperative complications, surgical trauma and healing time was decreased; operating time was reduced; costs were decreased.

ELIGIBILITY:
Inclusion Criteria:

* eyes requiring pars plana vitrectomy for various indications: such as dropped lens, intraocular blood, retinal detachments...etc.

Exclusion Criteria:

* patients who did not observed periodically during postoperative period.

Ages: 44 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were in the range 44 to 80 years, who had to undergo vitrectomy operation with different diagnosis were included in the study. Each participant had a complete ophthalmological examination which included best-corrected visual acuity (BCVA), slit lamp examination with and without pupil dilation, intraocular pressure (IOP) measurement with applanation tonometry and stereoscopic evaluation of the ocular fundus before decision of operation.
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
visual acuity

SECONDARY OUTCOMES:
postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ophthalmology,Hospital of Faculty of Medicine, Kocaeli University, Kocaeli, Turkey (Türkiye)